CLINICAL TRIAL: NCT00832403
Title: Gore Tex Implants in the Treatment of Atrophic Rhinitis
Acronym: RA
Status: Suspended | Type: Observational
Why Stopped: lack of new patients
Sponsor: Hospital Felicio Rocho (Other)
Responsible Party: Larissa Oliveira Lauriano, Hospital Felício Rocho
Other Study IDs: Rinite Atrófica cep/hfr
Record Dates: First submitted 2009-01-27; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Atrophic Rhinitis
Keywords: atrophic rhinitis; implants; Polytetrafluoroethylene
MeSH Terms: conditions — Rhinitis, Atrophic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- polytetrafluoroethylene
  Interventions: Other: implants of polytetrafluoroethylene in tha nasal fossa

INTERVENTIONS:
Other: implants of polytetrafluoroethylene in tha nasal fossa — surgical implants of polytetrafluoroethylene in the nasal fossa

SUMMARY:
This is a retrospective study, involving patients with atrophic rhinitis, that underwent Gore tex® implants in the nasal fossa.

The Fetid Rhinitis or Atrophic Ozena is a chronic illness characterized by yellowish secretion in the initial phase and the other phases with fetid crusts and atrophy of the mucous bone covering. Diverse theories exist that try to explain the appearance of this pathology, such as: hereditary factors, immunological alterations, viral infection and nutritional lack. Currently, its etiology remains unknown. As there isn't any ideal treatment already established, this technique improves the options of treatment.

All patients have improved after the procedure.

DETAILED DESCRIPTION:
Data about 5 patients that underwent surgery to implant polytetrafluoroethylene in the nasal fossa was collect. The symptoms and complications were described.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of atrophic rhinitis, with previous clinical treatment without good results

Exclusion Criteria:

* Patients with mental illness

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that were submit to surgery to treat atrophic rhinitis with implants in the nasal fossa.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
improvement of fetid crusts and atrophy of the mucous bone covering | after surgery recovery

SECONDARY OUTCOMES:
lack of side effects such as infection | after the treatment